CLINICAL TRIAL: NCT01020786
Title: Post-marketing Clinical Trial of Induction Chemotherapy of Pemetrexed Plus Carboplatin Followed by Pemetrexed Maintenance Therapy for Advanced Nonsquamous Non-small Cell Lung Cancer
Brief Title: A Study in Non-squamous Non Small Cell Lung Cancer in Asian Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12628; H3E-JE-JMII (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Carboplatin (Experimental): After four 21-day cycles of Pemetrexed plus Carboplatin treatment, Pemetrexed monotherapy is continued until study discontinuation.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Pemetrexed — Induction Therapy: 500 milligrams per square meter (mg/m^2) given intravenously (IV) on Day 1 of every 21-day cycle for 4 cycles.
  Maintenance Therapy: 500 mg/m^2 given IV on Day 1 of every 21-day cycle until disease progression or unacceptable toxicity.
  Other Names: Alimta; LY231514
Drug: Carboplatin — Dosage equal to area under the curve (AUC)6 milligrams per milliliter per minute (mg/mL/min) for participant, given IV on Day 1 of every 21-day cycle for 4 cycles.

SUMMARY:
To investigate efficacy and safety of the combination with pemetrexed plus carboplatin, followed by pemetrexed in patients with advanced nonsquamous Non Small Cell Lung Cancer (NSCLC) who receive at least one dose of the induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-squamous cell Non Small Cell Lung Cancer (NSCLC) disease
* Clinical stage IIIB/IV or recurrent disease after surgery
* No prior systemic chemotherapy, immunotherapy, targeted therapy or biological therapy, including adjuvant therapy
* Prior radiation therapy is allowed to less than 25% of the bone marrow
* Measurable disease as defined by response evaluation criteria in solid tumors (RECIST)
* The Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate organ function
* Estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* Clinically significant third-space fluid collections
* Central nervous system disease other than stable and treated brain metastasis
* More than 3 weeks interval between the surgery and enrollment request date
* Unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), for a 5 days period
* Unable or unwilling to take folic acid or vitamin B12 supplementation
* Unable to take corticosteroids.
* Serious concomitant disorder that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol
* Currently have and historically had interstitial pneumonitis (interstitial pneumonia) or pulmonary fibrosis manifested as opacity on Chest x-ray or Computed tomography (CT)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Japan (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi

REFERENCES:
- [Derived] Okamoto I, Aoe K, Kato T, Hosomi Y, Yokoyama A, Imamura F, Kiura K, Hirashima T, Nishio M, Nogami N, Okamoto H, Saka H, Yamamoto N, Yoshizuka N, Sekiguchi R, Kiyosawa K, Nakagawa K, Tamura T. Pemetrexed and carboplatin followed by pemetrexed maintenance therapy in chemo-naive patients with advanced nonsquamous non-small-cell lung cancer. Invest New Drugs. 2013 Oct;31(5):1275-82. doi: 10.1007/s10637-013-9941-z. Epub 2013 Mar 10. PMID 23475281

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Induction period: pemetrexed and carboplatin were administered for 4 cycles (1 cycle=21 days). Participants with documented complete response (CR), partial response (PR), or stable disease (SD) entered the maintenance therapy period (fifth cycle and after).
  Maintenance period: pemetrexed monotherapy until a discontinuation criterion was met.
Groups:
- Pemetrexed + Carboplatin: Induction therapy period (Pemetrexed + carboplatin): 500 milligrams per square meter (mg/m^2) of pemetrexed given intravenously (IV) on Day 1 of every 21-day cycle for 4 cycles.
  Carboplatin: dosage equal to the area under the curve (AUC) 6 milligrams per milliliter per minute (mg/mL/min) for participant, given IV on Day 1 of every 21-day cycle for 4 cycles.
  Maintenance therapy period (pemetrexed monotherapy): 500 mg/m^2 of pemetrexed given IV on Day 1 of every 21-day cycle until disease progression or unacceptable toxicity.
Period: Induction Period
Arm/Group | Pemetrexed + Carboplatin
Started | 109
Completed | 60 (Completed induction therapy. Completed=starting the maintenance therapy.)
Not Completed | 49
Not completed — Entry Criteria Not Met | 2
Not completed — Adverse Event | 10
Not completed — Progressive Disease | 31
Not completed — Investigator Decision | 3
Not completed — Withdrawal by Subject | 3
Period: Maintenance Period
Arm/Group | Pemetrexed + Carboplatin
Started | 60
Completed | 0
Not Completed | 60
Not completed — Adverse Event | 8
Not completed — Progressive Disease | 43
Not completed — Withdrawal by Subject | 8
Not completed — Sponsor Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 109
Age Continuous [Mean (Standard Deviation); unit: years] | 63.35 (8.692)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 69
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 109
Region of Enrollment [Number; unit: participants]
  Japan | 109
Percentage of Participants in Each Smoking Status Category at Study Entry [Number; unit: percentage of participants] — Percentage of participants in each category for smoking status. All of the percentages do not add up to 100% because of rounding.
  percentage of participants
    Current Smoker | 8.3
    Former Smoker | 61.5
    Never Smoker | 30.3
    Unknown | 0.0
Percentage of Participants in Each Histology Category [Number; unit: percentage of participants] — Percentage of participants in each of the following categories: adenocarcinoma, large cell lung carcinoma, and carcinoma, non-small cell, lung not otherwise specified (NOS).
  percentage of participants
    Adenocarcinoma Lung | 97.2
    Large Cell Lung Carcinoma | 2.8
    Carcinoma, Non-small Cell, Lung Not Otherwise S | 0
Percentage of Participants in Each Disease Stage [Number; unit: percentage of participants] — Percentage of participants in each disease stage category. Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body. Stage IIIB - cancer spread to opposite side of chest, more than 1 tumor within same lobe of lung; Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver. All of the percentages do not add up to 100% because of rounding.
  percentage of participants
    Stage IIIb | 30.3
    Stage IV | 66.1
    Other | 3.7
Percentage of Participants in Each Epidermal Growth Factor Receptor (EGFR) Mutation Status Category [Number; unit: percentage of participants] — Percentage of participants in each EGFR mutation status category.
  percentage of participants
    Positive | 22.0
    Negative | 57.8
    Unknown | 2.8
    Not Done | 17.4
Percentage of Participants in Each Eastern Cooperative Oncology Group (ECOG) Status [Number; unit: percentage of participants] — ECOG Performance Status (PS). Classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  0 - Fully Active
  1. - Ambulatory, Restricted Strenuous Activity
  2. - Ambulatory, No Work Activities
  3. - Partially Confined to Bed, Limited Self Care
  4. - Completely Disabled
  5. - Death
  percentage of participants
    0 - Fully Active | 33.9
    1 - Ambulatory, Restricted Strenuous Activity | 66.1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) During the Induction and Maintenance Therapy Periods
Description: PFS defined as time from enrollment date to first date of objective progression of disease or of death from any cause. Tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.0, which define when cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. Participants receiving any subsequent systemic anticancer therapy before objective progression or death were censored at date of last objective progression-free disease assessment before starting subsequent systemic anticancer therapy.
Time Frame: Enrollment to the date of progressive disease (PD) or the date of death from any cause (up to 18 months)
Population: Full Analysis Set (FAS): consists of the participants who received the induction combination therapy with pemetrexed and carboplatin; 31 participants were censored as they received subsequent systemic anticancer therapy before confirming objective PD or there was not a confirmed objective PD.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pemetrexed + Carboplatin: Induction therapy period (Pemetrexed + carboplatin): 500 milligrams per square meter (mg/m2) of pemetrexed given intravenously (IV) on Day 1 of every 21 day cycle for 4 cycles.
  Carboplatin: dosage equal to the area under the curve (AUC) 6 for participant, given IV on Day 1 of every 21 day cycle for 4 cycles.
  Maintenance therapy period (pemetrexed monotherapy): 500 mg/m2 of pemetrexed given IV on Day 1 of every 21 day cycle until disease progression or unacceptable toxicity.
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 109
months | 5.6 [4.3 to 7.2]

2. Secondary Outcome: Overall Survival (OS) During the Induction and Maintenance Therapy Periods
Description: OS was defined as the time from the enrollment date to the date of death from any cause. For participants who were alive, OS was censored at the last contact.
Time Frame: Enrollment to the date of death from any cause (up to 30.8 months)
Population: Full analysis set (FAS): consists of the participants who received the induction combination therapy with pemetrexed and carboplatin; 79 participants were censored as the observation period was not enough at the time of data cut-off for the primary endpoint (EP) of PFS. There were 48 participants censored at the final endpoint data cut-off.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 109
months
  Overall Survival (OS) at primary endpoint | NA [NA to NA] — The median and 95% confidence interval were not calculable because an insufficient number of participants reached the event at the time of the data cutoff.
  Overall Survival (OS) at final endpoint | 20.2 [16.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the time of final data cutoff.

3. Secondary Outcome: Percentage of Participants Who Achieve a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) During the Induction and Maintenance Therapy Periods
Description: Calculated as the percentage of participants who achieved a confirmed CR, PR, or SD. Tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.0, which define when cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. CR = disappearance of all target lesions. PR = 30% decrease in the sum of the longest diameter of target lesions. Progressive Disease (PD) = 20% increase in the sum of the longest diameter of target lesions. SD = small changes that do not meet above criteria.
Time Frame: Enrollment to date of progressive disease (up to 18 months)
Population: Full Analysis Set (FAS): consists of the participants who received the induction combination therapy with pemetrexed and carboplatin.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 109
percentage of participants
  CR+PR | 34.9 [26.0 to 44.6]
  CR+PR+SD | 72.5 [63.1 to 80.6]

4. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response (CR) or Partial Response (PR) During the Induction and Maintenance Therapy Periods
Description: Calculated as the percentage of participants who achieved a confirmed CR or PR. Tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.0, which define when cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. CR = disappearance of all target lesions. PR = 30% decrease in the sum of the longest diameter of target lesions. Progressive Disease (PD) = 20% increase in the sum of the longest diameter of target lesions. Stable Disease (SD) = small changes that do not meet above criteria.
Time Frame: Enrollment to date of progressive disease (up to 18 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 109
percentage of participants
  CR | 0.0
  PR | 34.9

5. Secondary Outcome: Progression Free Survival (PFS) During the Maintenance Therapy Period
Description: Measured from the date of the first dose of the maintenance therapy. Calculated by subtracting induction therapy period from PFS. Tumor response assessed using Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.0; define when cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. Participants receiving any subsequent systemic anticancer therapy before objective progression or death were censored at date of last objective progression-free disease assessment before starting subsequent systemic anticancer therapy.
Time Frame: From the start of maintenance therapy in Cycle 5 (21-day cycle) until the date of measured progressive disease (PD) or death from any cause (up to 24.4 months)
Population: Analysis set: Maintenance-treated participants who received maintenance therapy with pemetrexed; 20 and 12 participants were censored at time of primary endpoint (18 months) and final endpoint. They received subsequent systemic anticancer therapy before confirming objective PD or there was not a confirmed objective PD at cut-off.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 60
months
  PFS at primary endpoint | 3.9 [2.8 to 5.0]
  PFS at final endpoint | 3.9 [3.2 to 5.2]

6. Secondary Outcome: Overall Survival (OS) During the Maintenance Therapy Period
Description: OS was defined as the duration from the date of the first dose of the maintenance therapy to the date of death from any cause and was calculated by subtracting the induction therapy period from OS. Participants receiving any subsequent systemic anticancer therapy before objective progression or death were censored at date of last objective progression-free disease assessment before starting subsequent systemic anticancer therapy. For participants who were alive, OS was censored at the last contact.
Time Frame: From the start of maintenance therapy in Cycle 5 (21-day cycle) until the date of measured progressive disease (PD) or death from any cause (up to 26.3 months)
Population: Analysis set: Maintenance-treated participants, which consist of the participants who received the maintenance therapy with pemetrexed; 56 participants and 38 participants were censored as the observation period was not enough at the time of data cut-off for the primary endpoint, PFS, and final endpoint, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 60
months
  Overall Survival (OS) at primary endpoint | NA [NA to NA] — The median and the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the time of the 2-year data cutoff.
  Overall Survival (OS) at final endpoint | NA [21.0 to NA] — The median and the upper 95% confidence interval were not calculable because an insufficient number of participants reached the event at the time of final data cutoff.

7. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) During the Maintenance Therapy Period
Description: Percentage of participants who achieved confirmed CR (disappearance of all target lesions), PR (30% decrease in sum of longest diameter of target lesions), or SD (small changes that do not meet above criteria). Response derived from target lesion assessments performed before maintenance therapy (as baseline), during maintenance therapy (as post-baseline), and non-target lesion assessments performed during maintenance therapy according to RECIST guideline version 1.0, defines when cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments.
Time Frame: From the start of maintenance therapy in Cycle 5 (21-day cycle) until the date of measured progressive disease (PD) or death from any cause (up to 18 months)
Population: Analysis set: Maintenance-treated participants, which consist of the participants who received the maintenance therapy with pemetrexed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 60
percentage of participants
  CR+PR | 3.3 [0.4 to 11.5]
  CR+PR+SD | 48.3 [35.2 to 61.6]

8. Secondary Outcome: Percentage of Participants Who Observe a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) During the Induction Therapy Period
Description: Calculated as the percentage of participants who achieved a CR, PR, or SD (confirmed or not). Tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.0, which define when cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. CR = disappearance of all target lesions. PR = 30% decrease in the sum of the longest diameter of target lesions. Progressive Disease (PD) = 20% increase in the sum of the longest diameter of target lesions. SD = small changes that do not meet above criteria.
Time Frame: Enrollment to the date of PD, or end of induction period up to Cycle 4 (21-day cycle)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 109
percentage of participants | 81.7 [73.1 to 88.4]

9. Secondary Outcome: Percentage of Participants Who Achieve a Complete Response (CR) or a Partial Response (PR) During the Induction Therapy Period
Description: Calculated as percentage of participants who achieved a CR or PR (confirmed or not). Tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.0, which define when cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. CR = disappearance of all target lesions. PR = 30% decrease in sum of the longest diameter of target lesions. Progressive Disease (PD) = 20% increase in the sum of longest diameter of target lesions. Stable Disease (SD) = small changes that do not meet above criteria.
Time Frame: Enrollment to date of PD, or end of induction period up to Cycle 4 (21-day cycle)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 109
percentage of participants | 38.5 [29.4 to 48.3]

ADVERSE EVENTS:
Time Frame: Treatment period plus 30 day follow-up period (up to 30.8 months)
Description: Adverse events were updated to add the adverse events occurring after the data cut-off date for the primary endpoint (PFS) to those events previously reported.
Arm/Group | Pemetrexed + Carboplatin
Serious Adverse Events (participants affected / at risk) | 17/109
Other Adverse Events (participants affected / at risk) | 109/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin (N=109)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Obstruction (General disorders) | 1 (1)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin (N=109)
Anaemia (Blood and lymphatic system disorders) | 47 (59)
Leukopenia (Blood and lymphatic system disorders) | 44 (147)
Lymphopenia (Blood and lymphatic system disorders) | 14 (23)
Neutropenia (Blood and lymphatic system disorders) | 58 (193)
Thrombocytopenia (Blood and lymphatic system disorders) | 30 (84)
Abdominal pain (Gastrointestinal disorders) | 9 (15)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Cheilitis (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 52 (110)
Diarrhoea (Gastrointestinal disorders) | 25 (37)
Nausea (Gastrointestinal disorders) | 81 (206)
Stomatitis (Gastrointestinal disorders) | 22 (27)
Vomiting (Gastrointestinal disorders) | 46 (71)
Fatigue (General disorders) | 75 (181)
Influenza like illness (General disorders) | 7 (8)
Injection site reaction (General disorders) | 10 (10)
Malaise (General disorders) | 12 (19)
Oedema (General disorders) | 8 (8)
Pyrexia (General disorders) | 35 (56)
Nasopharyngitis (Infections and infestations) | 7 (10)
Pneumonia (Infections and infestations) | 10 (12)
Alanine aminotransferase increased (Investigations) | 62 (152)
Aspartate aminotransferase increased (Investigations) | 60 (153)
Blood albumin decreased (Investigations) | 15 (19)
Blood alkaline phosphatase increased (Investigations) | 20 (23)
Blood bilirubin increased (Investigations) | 7 (12)
Blood calcium decreased (Investigations) | 11 (17)
Blood creatinine increased (Investigations) | 9 (17)
Blood lactate dehydrogenase increased (Investigations) | 38 (72)
Blood potassium increased (Investigations) | 7 (11)
Blood sodium decreased (Investigations) | 7 (15)
Blood urea increased (Investigations) | 10 (16)
Gamma-glutamyltransferase increased (Investigations) | 31 (42)
Haemoglobin decreased (Investigations) | 52 (79)
Neutrophil count decreased (Investigations) | 30 (98)
Platelet count decreased (Investigations) | 65 (225)
Red blood cell count decreased (Investigations) | 8 (8)
Weight decreased (Investigations) | 11 (15)
White blood cell count decreased (Investigations) | 42 (131)
Decreased appetite (Metabolism and nutrition disorders) | 82 (199)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Dizziness (Nervous system disorders) | 20 (27)
Dysgeusia (Nervous system disorders) | 11 (13)
Headache (Nervous system disorders) | 15 (20)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (12)
Insomnia (Psychiatric disorders) | 23 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 17 (34)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (12)
Rash (Skin and subcutaneous tissue disorders) | 37 (50)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days